CLINICAL TRIAL: NCT03181126
Title: A Phase 1 Dose Escalation, Open-Label Study of Venetoclax in Combination With Navitoclax and Chemotherapy in Subjects With Relapsed/Refractory Acute Lymphoblastic Leukemia or Relapsed/Refractory Lymphoblastic Lymphoma
Brief Title: A Study of Venetoclax in Combination With Navitoclax and Chemotherapy in Subjects With Relapsed/Refractory Acute Lymphoblastic Leukemia or Relapsed/Refractory Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-106
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Lymphoblastic Lymphoma
Keywords: Relapsed of Refractory Acute Lymphoblastic Leukemia; Cancer; Venetoclax; Navitoclax
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — navitoclax; Drug Therapy; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Navitoclax + Chemotherapy (Experimental): Venetoclax weight-adjusted doses administered orally every day (QD) starting on Day 1 + navitoclax various, weight-adjusted doses administered orally QD starting on Day 3 + chemotherapy (peg-asparaginase [or any other forms of asparaginase], vincristine, dexamethasone) and tyrosine kinase inhibitor [TKI, if applicable]). This regimen and any of its components may be delayed, reduced or omitted at the discretion of the Investigator.
  Interventions: Drug: Navitoclax; Drug: Chemotherapy; Drug: Venetoclax

INTERVENTIONS:
Drug: Navitoclax — tablet
  Other Names: ABT-263
Drug: Chemotherapy — peg-asparaginase (or other form of asparaginase, per local standard of care (intravenous) + vincristine (intravenous) + dexamethasone (oral) + tyrosine kinase inhibitor (TKI) (if applicable, oral)
Drug: Venetoclax — tablet
  Other Names: ABT-199 GDC-0199

SUMMARY:
This dose-escalating study is to determine the safety, pharmacokinetics, and preliminary efficacy of venetoclax in combination with navitoclax and chemotherapy in adult and pediatric participants with relapsed/refractory acute lymphoblastic leukemia (ALL) or relapsed/refractory lymphoblastic lymphoma. A safety expansion cohort of approximately 20 patients may be enrolled in addition to the 50 participants in dose-escalation cohort.

ELIGIBILITY:
Inclusion Criteria:

* Must have relapsed or refractory acute lymphoblastic leukemia (ALL) or relapsed or refractory lymphoblastic lymphoma (LL). Refractory is defined as persistent disease after at least 2 courses of chemotherapy.

  * Participants with ALL with Philadelphia chromosome or with an ABL class targetable fusion are eligible.
  * Participants with LL must have radiographic evidence of disease
* Participants <= 18 years of age who do not have a standard of care treatment option available.
* Must weigh greater than or equal to 20 kg.
* Must be able to swallow pills.
* Must have adequate hepatic and kidney function.
* Must have adequate performance status:

  * Participants less than or equal to 16 years of age: Lansky greater than or equal to 50
  * Participants greater than 16 years of age: Karnofsky greater than or equal to 50 or Eastern Cooperative Oncology Group (ECOG) less than 3.

Exclusion Criteria:

* Participant has central nervous system (CNS) disease with cranial involvement that requires radiation.
* Participants who are less than 100 days post-transplant, or greater than 100 days post-transplant with active graft versus host disease (GVHD), or are still continuing post-transplant immunosuppressant therapy within 7 days prior to the first dose of study drug.
* Participants who have received any of the following prior to the first dose of study drug:

  * Inotuzumab within 30 days (if participant received inotuzumab > 30 days prior to Day 1, must have ALT, AST and bilirubin < ULN).
  * A biologic agent (i.e., monoclonal antibodies) for anti-neoplastic intent within 30 days
  * CAR-T infusion or other cellular therapy within 30 days
  * Any anti-cancer therapy including blinatumomab, chemotherapy, radiation therapy targeted small molecule agents or investigational agents within 14 days, or 5 half-lives, whichever is shorter

    * Exception: Philadelphia Chromosome (Ph)+ ALL subjects on TKIs at Screening may enroll and remain on Tyrosine Kinase Inhibitor (TKI) therapy to control disease. Participants on venetoclax at screening may enroll and remain on venetoclax.
  * Steroid therapy for anti-neoplastic intent within 5 days
  * Hydroxyurea that is ongoing (hydroxyurea is permitted up to the first dose)
  * A strong or moderate CYP3A inhibitor or inducer within 7 days
  * Aspirin within 7 days, or 5 half-lives, whichever is longer
  * An excluded antiplatelet/anticoagulant drug or a herbal supplement that affects platelet function within 7 days, or 5 half-lives, whichever is longer
* Participants with malabsorption syndrome or any other condition that precludes enteral administration.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Cmax of Venetoclax + Navitoclax | Up to approximately 9 months
  Maximum observed plasma concentration (Cmax) of venetoclax + navitoclax
AUC of Venetoclax + Navitoclax | Up to approximately 9 months
  Area under the plasma concentration-time curve (AUC) of venetoclax + navitoclax
Tmax of Venetoclax + Navitoclax | Up to approximately 9 months
  Time to Cmax (Tmax) of Venetoclax + Navitoclax
CL/F of Venetoclax + Navitoclax | Up to approximately 9 months
  Apparent oral clearance (CL/F) of venetoclax + navitoclax
Number of participants with dose-limiting toxicities (DLT) | Up to approximately 28 days after initial dose of study drug
  A DLT is any Grade 3 or higher non-hematologic adverse event (AE) with exceptions outlined in the protocol. AEs and toxicities that occur beyond the DLT assessment period will also be evaluated by the investigator and AbbVie and may be considered as dose-limiting.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 9 months after the last subject has enrolled into the study
  PFS is defined as the number of days from the date of enrollment to the date of earliest disease progression or death.
Partial Response (PR) rate | Up to 9 months after the last subject has enrolled into the study
  PR defined as no peripheral blasts or peripheral blood absolute blast count decreased by ≥ 50% from baseline, bone marrow with 5 - 25% blasts and at least a 50% decrease in bone marrow blast percent from baseline, no evidence of extramedullary disease.
Number of Participant who Proceed to Stem Cell Transplantation or Chimeric antigen receptor T-cell (CAR-T) Therapy | Up to 9 months after the last subject has enrolled into the study
  Determine the number of participants who proceed to stem cell transplantation or CAR-T therapy.
Overall survival (OS) | Up to 9 months after the last subject has enrolled into the study
  OS is defined as the number of days from the date of enrollment to the date of death.
Objective response rate (ORR) | Up to 9 months after the last subject has enrolled into the study
  The proportion of subjects with objective response rate (complete response [CR] + CR incomplete recovery [CRi] + CR without platelet recovery [CRp]) for ALL subjects and (CR+PR) for LL subjects.
Complete Response (CR) rate | Up to 9 months after the last subject has enrolled into the study
  CR defined as hematologic recovery (absolute neutrophil count [ANC] greater than or equal to 500/μL; platelet counts greater than or equal to 75,000/μL), evidence of trilineage hematopoiesis in the bone marrow and less than 5% blasts in the bone marrow, absence of circulating blasts, and no evidence of extramedullary disease.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (15):
- United States (12):
  - City of Hope /ID# 169029, Duarte, California
  - LPCH Stanford /ID# 163337, Palo Alto, California
  - University of Chicago /ID# 163369, Chicago, Illinois
  - Washington University-School of Medicine /ID# 165689, St Louis, Missouri
  - Univ NC Chapel Hill /ID# 163509, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital /ID# 164619, Cincinnati, Ohio
  - Nationwide Childrens Hospital /ID# 163372, Columbus, Ohio
  - Oregon Health and Science University /ID# 165690, Portland, Oregon
  - St Jude Children's Research Hospital /ID# 163335, Memphis, Tennessee
  - UT Southwestern Medical Center /ID# 163346, Dallas, Texas
  - MD Anderson Cancer Center at Texas Medical Center /ID# 163327, Houston, Texas
  - University of Wisconsin-Madiso /ID# 165691, Madison, Wisconsin
- Australia (3):
  - Alfred Hospital /ID# 169576, Melbourne, Victoria
  - Victorian Comprehensive Cancer /ID# 165710, Melbourne, Victoria
  - Royal Children's Hospital /ID# 163322, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Badawi M, Gopalakrishnan S, Engelhardt B, Palenski T, Karol SE, Rubnitz JE, Menon R, Salem AH. Dosing of Venetoclax in Pediatric Patients with Relapsed Acute Myeloid Leukemia: Analysis of Developmental Pharmacokinetics and Exposure-Response Relationships. Clin Ther. 2024 Oct;46(10):759-767. doi: 10.1016/j.clinthera.2024.09.008. Epub 2024 Oct 5. PMID 39368878
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/venetoclax_M16-106.pdf